CLINICAL TRIAL: NCT05474222
Title: Horizon Eagle Fatherhood Program
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Horizon Outreach (Other)
Responsible Party: Principal Investigator, Michael Young, Principal Investigator, Horizon Outreach
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2022-06-11; First posted 2022-07-26 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Responsible Fatherhood Programming

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned, in a three to one ratio, to the intervention group, or the control group. All participants will complete a pretest questionnaire and have access to case management services. The intervention group will receive 40 hours of classroom instruction, then all participants will complete a posttest questionnaire. Following the posttest all participants will have access to workforce training. Six months after the posttest, all participants will complete a follow-up questionnaire.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Horizon Eagle Fatherhood Programming - classroom instruction (Experimental): The intervention (the Horizon Eagle Fatherhood Programming) is an intensive 40-hour classroom-based program taught by project staff. This instruction addresses topics such as Fatherhood Development, Relationship Enhancement, and Financial Literacy, and features the 24/7 Dad curriculum as part of the instruction. Intervention participants and control participants will have an opportunity to participate in case management services and workforce training.
  Interventions: Other: Horizon Eagle Fatherhood Program - classroom instruction
- Control (No Intervention): The control group does not receive any part of the classroom instruction that the intervention group receives. Like the intervention group, however, the control group does have access to case management and workforce training.

INTERVENTIONS:
Other: Horizon Eagle Fatherhood Program - classroom instruction — The intervention group (the Horizon Eagle Fatherhood Programming) receives 40 hours of classroom instruction
  Arms: Horizon Eagle Fatherhood Programming - classroom instruction

SUMMARY:
Horizon Outreach has developed the Horizon Eagle Fatherhood Program (HEFP). HEFP includes a program/services aspect, but also includes a rigorous evaluation component, featuring a randomized control trial (RCT) research design. The evaluation will determine the effect of the Horizon Eagle Fatherhood Program with fathers aged 18 and up in Houston, Texas. Specifically, the research is examining the effects of the program relative to: (1) improvement in healthy relationship and marriage skills, (2) improvement in parenting skills, (3) improvement in conflict resolution and anger management skills, and (4) improvement in financial management skills and progress toward greater economic stability.

Program participants will be randomly assigned to either the intervention group or the control group. Participants assigned to the intervention group will receive the program now. Participants assigned to the control group will have an opportunity to receive the program later. All participants (intervention and control) will complete a pretest questionnaire. Intervention participants will then participate in the Horizon Eagle Fatherhood program. This is an intensive 40-hour classroom-based program taught by project staff. Both intervention and control participants will receive case management services. Following completion of the program by the intervention participants, all participants will complete a posttest questionnaire. After completion of the posttest, all participants will have an opportunity to participate in a workforce training program. Six months following posttest, all participants will complete a third questionnaire. In addition, a selected number of participants will participate in focus groups. After completing the six-month follow-up questionnaire, participants from the control group may participate in the 40 hours of classroom instruction, should they choose to do so.

This RCT research design component of the Horizon Eagle Fatherhood Program began in June of the second project year. Prior to the start of the RCT, a pilot/readiness project with no control group was conducted. This was followed by a short-term pilot of the RCT.

DETAILED DESCRIPTION:
Horizon Outreach has developed the Horizon Eagle Fatherhood Program (HEFP). HEFP includes a program/services aspect, but also includes a rigorous evaluation component, featuring a randomized control trial (RCT) research design. The evaluation will determine the effect of the Horizon Eagle Fatherhood Program with fathers aged 18 and up in Houston, Texas. Specifically, the research is examining the effects of the program relative to: (1) improvement in healthy relationship and marriage skills, (2) improvement in parenting skills, (3) improvement in conflict resolution and anger management skills, and (4) improvement in financial management skills and progress toward greater economic stability.

The intervention includes 40 hours of classroom instruction. This instruction addresses topics such as Fatherhood Development, Relationship Enhancement, and Financial Literacy, and features the 24/7 Dad curriculum as part of the instruction. All participants will have the opportunity to participate in enhanced case management, and workforce training. Thus, the evaluation will determine whether the classroom instruction component makes a difference in outcome variables, over and above any difference that may be made bu the case management and workforce training.

Program participants will be randomly assigned to either the intervention group or the control group. Participants assigned to the intervention group will receive the program now. Participants assigned to the control group will have an opportunity to receive the program later. All participants (intervention and control) will complete a pretest questionnaire. Intervention participants will then participate in the Horizon Eagle Fatherhood program. This is an intensive 40-hour classroom-based program taught by project staff. Both intervention and control participants will receive case management services. Following completion of the program by the intervention participants, all participants will complete a posttest questionnaire. After completion of the posttest, all participants will have an opportunity to participate in a workforce training program. Six months following posttest, all participants will complete a third questionnaire. In addition, a selected number of participants will participate in focus groups. After completing the six-month follow-up questionnaire, participants from the control group may participate in the 40 hours of classroom instruction, should they choose to do so.

There are four primary research questions. Does the Horizon Eagle intervention produce improvement in (1) Healthy relationship and marriage skills? (2) Parenting skills? (3) Conflict resolution and anger management skills? (4) Financial management and progress toward economic stability? Participants will be randomly assigned, in a 3:1 ratio, to treatment or control conditions. All control participants who complete a pretest questionnaire, posttest questionnaire, and/or a follow-up questionnaire will be included in the data analysis. For participants in the intervention group, those who complete at least a portion of the intervention, will be included in the analysis. The analysis will determine whether those participants who the investigators assigned to the intervention group, and who completed at least a portion of the intervention, improved in self-reported attitudes and behaviors, when compared to participants in the control condition.

The program requires that written participant consent be obtained before participation in the program and prior to the collection of any data. Participants will be informed of the study the first time they meet with the intake coordinator. Prior to beginning the intake process, participants will be provided with a detailed informed consent form explaining the aims of the program, benefits, and any potential risk of the program (see Appendix). Risk within this project is identified as minimal. Participants may feel uncomfortable responding to some of the questions in the questionnaire, as it may bring up topics of conversation related to relationships and family communication. Participants will be informed that responses to questions are voluntary. Participants will be informed of the benefits of the program, including strengthening family relationships and bonding, and improvement in communication skills. Participants who have provided written consent to participate in the project (and who are at least 18) will complete the pre-test questionnaire (baseline) in an appropriate setting, at the intake. The pre-test questionnaire will be completed before the implementation of the intervention curricula.

Fathers who have provided written consent to participate in the project will complete the questionnaire in an appropriate setting, prior to program implementation. The questionnaire will have items to measure the major outcomes of the project at baseline. The evaluation team will train project staff in evaluation procedures, by recruiting a Data Collection Specialist (DCS) to train with specific attention to questionnaire administration and data collection protocols. The DCS and Intake Coordinator will distribute a tablet to each subject in the administration setting. The DCS or Intake Coordinator will input the following for each subject's questionnaire: the subject number and test time (pre-test, post-test, or follow-up). The subject code number will be the same number for all three questionnaires, thus allowing us to match subjects' initial questionnaire responses with responses across administrations.

To maximize the validity of these self-report data, the DCS will emphasize that (a) all individual responses are confidential and will not be revealed to family members, or law enforcement officials, (b) participants are to keep their eyes on their own questionnaire and not to discuss any of the questions with other participants while completing the questionnaire, and (c) participants will be told they have the right to "pass" on any question they do not wish to answer. They will, however, be encouraged to answer all questions, with emphasis placed on the importance of honest answers.

Research participants will complete all questionnaires via Qualtrics web-based software. Participants will use the tablets to connect with Qualtrics using a wireless Internet connection. To make sure there are minimal problems with questionnaire completion and submission, the DCS will use a tablet to demonstrate how to answer questions, move to the next page of the questionnaire and how to submit the completed questionnaire. Qualtrics software is cloud-based and can be connected to with wireless internet connectivity. All information collected will use a secure and encrypted wireless connection.

To examine longitudinal changes in outcome variables, analysis of covariance will be used. The pretest score for the variable under consideration will be used as a covariate, other covariates will also include any demographic variable for which the intervention and control group differ at pretest. For all analyses, the Bonferroni procedure for alpha correction will be used when conducting multiple comparisons, to guard against inflated Type I error.

ELIGIBILITY:
Inclusion Criteria:

* Must be a father
* At least 18 years of age
* At least one child under the age of 24.

Exclusion Criteria:

* Not a father
* Not at least 18 years of age
* No children under the age of 24.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Eligibility is based on self-representation of gender identity.
Enrollment: 1200 (Estimated)
Dates: Start 2022-07-05 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Improvement in healthy marriage/relationship communication skills scores | Pretest to Follow-up (six months after completion of the intervention - about 7 months after the pretest)
  This outcome is the participants' score on a healthy marriage/relationship skills scale. This is a 10 item scale. It was used in an article recently published in Family Relations. The principal investigator for the present study (Young) was also the lead author for the study published in Family Relations. A sample item from the scale is "It is important to show appreciation for others." In the Family Relations study the items in the scale loaded on a single factor at .56 or above. The internal consistency (Chronbach's alpha) at pretest was .87. The percentage of the variance explained by the first component was 46. The results table will report the mean scores of the intervention and control groups at pretest, posttest and follow-up, as well as the results from the statistical analysis.
Improvement in conflict management/resolution skills scores | Pretest to Follow-up (six months after completion of the intervention - about 7 months after the pretest)
  This outcome is the participants' score on a conflict management/ resolution skills scale. This is a 6 item scale. It was used in an article recently published in Family Relations. The principal investigator for the present study (Young) was also the lead author for the study published in Family Relations. A sample item from the scale is "I follow through on promises and agreements." In the Family Relations study the items in the scale loaded on a single factor at .60 or above. The internal consistency (Chronbach's alpha) at pretest was .83. The percentage of the variance explained by the first component was 54.The results table will report the mean scores of the intervention and control groups at pretest, posttest and follow-up, as well as the results from the statistical analysis.
Improvement in attitudes about personal finances scores | Pretest to Follow-up (six months after completion of the intervention - about 7 months after the pretest)
  This outcome is the participants' score on an attitudes about personal finances scale. This is a 6 item scale. It was used in an article recently published in Family Relations. The principal investigator for the present study (Young) was also the lead author for the study published in Family Relations. A sample item from the scale is "I can reduce conflict about money through discussion and problem solving." In the Family Relations study the items in the scale loaded on a single factor at .63 or above. The internal consistency (Chronbach's alpha) at pretest was .72 and .94 at posttest.The results table will report the mean scores of the intervention and control groups at pretest, posttest and follow-up, as well as the results from the statistical analysis.
Improvement in job/career skills score | Pretest to Follow-up (six months after completion of the intervention - about 7 months after the pretest)
  This outcome is the participants' score on a job/career skills scale. This is a 6 item scale. It has been used in previous evaluations, including the final impact report (Fluegeman, S. Hernandez, A. Young, M. 2020) examining the Impact Evaluation of the Brothers United Fatherhood Program in Toledo, Ohio. This evaluation was conducted by Educational Evaluators, Inc. A sample item from the scale is "I feel confident in my ability to conduct an effective job search for a job I want." Internal consistency, measured by Cronbach's alpha, using the six items comprising the measure, were .72 at pretest and .94 at posttest in the Brothers United study. The principal investigator for the present study (Young) was also a co-author for the Brothers United study. The results table will report the mean scores of the intervention and control groups at pretest, posttest and follow-up, as well as the results from the statistical analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Young, Ph.D., Principal Investigator — Educational Evaluators, Inc; Center for Evidence-Based Programming
Locations (1):
- Horizon Outreach, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided
Yes - The funding agency, Office of Family Assistance (OFA), may require that data be archived so that other researchers may have access. We will comply with whatever OFA asks us to do.